CLINICAL TRIAL: NCT06941831
Title: Testing an mHealth Digital Dashboard to Improve Quality of Delivery of Evidence-based Interventions That Promote Family Mental Health and Functioning in Rwanda: A Hybrid Type 3 Study
Brief Title: Rwanda Digital Dashboard Hybrid Type 3 Implementation Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 5116621; R01MH136200 (NIH)
Record Dates: First submitted 2025-04-11; First posted 2025-04-24 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: IPV; Mental Health; Discipline Practices; Quality Assurance; Provider Confidence; Provider Skill; Quality of Life
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care Sugira Muryango Implementation (Active Comparator): Sugira Muryango delivery using usual care data entry, supervision, and quality monitoring tools and protocols (paper forms, static data entry platform).
  Sugira Muryango is a home-visiting intervention that promotes playful parenting, father engagement, improved nutrition, care seeking, and family functioning to promote ECD, positive parent-child relationships, and healthy child development. Sugira Muryango integrates these core components into 12 modules and two booster/follow-up sessions (3 and 6-months after intervention).
  Interventions: Other: Usual Care - Sugira Muryango Implementation
- Digital Dashboard Supported (Experimental): Sugira Muryango delivery using a Digital dashboard aimed at improving data collection, monitoring, and usability, facilitating social services referrals, and interventionist supervision and training.
  Sugira Muryango is a home-visiting intervention that promotes playful parenting, father engagement, improved nutrition, care seeking, and family functioning to promote ECD, positive parent-child relationships, and healthy child development. Sugira Muryango integrates these core components into 12 modules and two booster/follow-up sessions (3 and 6-months after intervention).
  Interventions: Other: Digital Dashboard-Supported Sugira Muryango Implementation

INTERVENTIONS:
Other: Digital Dashboard-Supported Sugira Muryango Implementation — Arm investigating technology-supported delivery of Sugira Muryango, specifically, the use of a Digital Dashboard tool developed in partnership with the University of Rwanda. Developed using co-design and user interface/user experience techniques, the Dashboard (a) streamlines collection of data on evidence-based intervention quality and reach; (b) improves visibility and searchability of implementation data by region; (c) facilitates caregiver mental health and social services referrals and follow up, and (d) serves as a training platform with resources to enhance lay worker fidelity (content-specific skills) and competence (cross-cutting skills) in evidence-based intervention delivery.
  Arms: Digital Dashboard Supported
Other: Usual Care - Sugira Muryango Implementation — Sugira Muryango intervention is delivered using traditional supervision, data entry, and quality monitoring tools.
  Arms: Usual Care Sugira Muryango Implementation

SUMMARY:
Mental disorders are leading causes of the health-related burden globally, and in Rwanda the intergenerational mental health consequences of the 1994 Genocide against the Tutsi persist and are further compounded by poverty, such that recent studies have found 20% of the Rwandan population has one or more mental disorders.

The Research Program on Children and Adversity (RPCA) has expanded its evidence-based home-visiting Sugira Muryango (SM) in Rwanda. The current study aims to assess a digitally enhanced delivery of Sugira Muryango to meet the needs of the Government of Rwanda in expanding the mental health and social services infrastructure.

The proposed research will test the feasibility, acceptability and impact of a technology-enabled service delivery model using a digital tool that streamlines data collection, improves visibility of key program performance metrics, and serves as a resource for learning materials that can be used for continuous learning and training of a non-specialized workforce that is delivering an evidence-based intervention that improves caregiver mental health and family functioning. What the team learn from technology-supported delivery of Sugira Muryango - an evidence-based, trauma-informed, family-based behavioral intervention in Rwanda - can be used to improve the efficiency, effectiveness, and scalability of evidence-based mental health services in Rwanda and globally.

DETAILED DESCRIPTION:
Globally, mental disorders are the second largest contributor to the burden of disease in adults. In settings disrupted by war and civil unrest, violence and loss contribute to significant unaddressed burden of mental disorders and family violence in adults with subsequent risks to children. In Rwanda the intergenerational mental health consequences of the 1994 Genocide against the Tutsi in Rwanda persist; recent studies found that 20% of the Rwandan population has one or more mental disorders with the highest rates observed in Genocide survivors.

Sugira Muryango is an evidence-based, trauma-informed, family-based behavioral intervention to promote healthy family functioning, early childhood development and reduce family violence. In several trials, Sugira Muryango has led to improvements in parental mental health and child development outcomes including social and emotional development of children, improved caregiver mental health and reductions in family violence. To support scaling the intervention the University of Rwanda and other partners developed a Digital Dashboard tool that: (a) streamlines collection of data on evidence-based intervention quality and reach; (b) improves visibility and searchability of implementation data by region; (c) facilitates caregiver mental health and social services referrals and follow up; and (d) serves as a training platform with resources to enhance interventionist fidelity and competence. In the context of understanding important factors for scaling evidence-based interventions, the proposed research will investigate dashboard-supported delivery of Sugira Muryango in terms of its reach, efficiency, and cost effectiveness.

This Hybrid Type 3 implementation-effectiveness study will collect outcomes measuring the program's effectiveness, quality of program delivery, feasibility, and acceptability from program beneficiaries, the interventionists, the interventionists' supervisors, and community stakeholders.

The study will compare the trajectories of fidelity, competence, and self-efficacy between dashboard-supported delivery and standard delivery. The study will also include social network analysis to understand how the characteristics of networks comprised of supervisors and interventionists affect trajectories over time. Lastly, the study will investigate the impact of dashboard-supported delivery by comparing the difference in child and caregiver mental health outcomes with standard delivery. These data will be used to analyze cost-effectiveness and return on investment of the intervention as delivered with and without the Dashboard. The results of the proposed research will identify scalable pathways to accelerate integration of technology and evidence-based mental health services into policy and practice in Rwanda.

Specific study aims and hypotheses are listed below:

Aim 1: Conduct a Hybrid Type 3 implementation-effectiveness cluster randomized trial to compare Dashboard-supported delivery of Sugira Muryango to standard delivery in Kirehe District (12 sectors).

* Aim 1.1: Compare competence and fidelity of IZUs' Sugira Muryango technology-enabled delivery compared to standard delivery.
* Hypothesis 1.1: IZU competence and fidelity scores for Dashboard-supported delivery will be superior to standard delivery.
* Aim 1:2: Investigate whether Dashboard-supported delivery affects IZU sustainment of evidence-based practices.
* Hypothesis 1.2: Dashboard-supported delivery will improve IZU readiness to change and buy-in thereby moderating adoption and sustainment of evidence-based practices.

Aim 2: Use social network analysis to examine cross-site learning-communications, knowledge flow, stakeholder interactions-across the PLAY Collaborative. The investigative team will compare sectors with and without Dashboard-supported delivery in Kirehe District.

* Aim 2.1: Compare the structure of communication and knowledge networks between Dashboard-supported and standard delivery by examining key metrics of network size, density, and centrality.
* Hypothesis 2.1: Technology-supported compared to standard delivery will have higher cross-site learning that is manifest in larger network size, density, and centrality measures.
* Aim 2.2: Examine effects of supervisors' personal networks characteristics (network size, communication frequency, quality and content of interactions) on IZU fidelity, competence, and knowledge of mental health promotion.
* Hypothesis 2.2: Personal network characteristics for supervisors (egos) and IZUs (alters/peers) will improve IZUs' competence, fidelity, internalized mental health knowledge, and self-efficacy.

Aim 3: Leverage GoR infrastructure to examine whether technology-supported delivery increases Sugira Muryango impact, efficiency, and return-on-investment. Child and caregiver behavioral, child development, and family violence outcomes will be used to conduct incremental cost-effectiveness and return on investment analyses that evaluate benefits from a societal perspective.

* Hypothesis 3.1: Dashboard-supported delivery will have superior effects on mental health, family violence, and child development outcomes compared with standard delivery.
* Hypothesis 3.2: Dashboard-supported delivery will demonstrate greater efficiency (e.g., time-to-resolution of risk-of-harm cases of family mental health and violence). - Hypothesis 3.3: Technology-supported delivery will be cost-effective and provide value based on social returns criteria.

ELIGIBILITY:
Inclusion Criteria:

* Household inclusion criteria: Participants must be the primary caregiver to a child between birth and 36 months. Caregivers must live in the same household as the child and must be the child's legal guardian. Legal guardians may be parents, aunts, uncles, grandparents, or foster parents. Participants must be categorized as Ubudehe 1 under the socio-economic categorization of households from LODA.
* Government Official inclusion criteria: Government officials must be located at the Village, Cell, Sector and/or District level and must participate in the 1-day ECD training. Government officials must also agree to participate in the PLAY Collaborative activities throughout the course of program delivery.
* IZU interventionist inclusion criteria: IZUs must be a part of the Inshuti z'Umuryango/Friends of the Family program, must be over the age of 18, and must be literate in Kinyarwanda.
* Cell Level IZU Mentor inclusion criteria: Cell Level IZU Coordinators must be situated at the Cell Level and able to supervise at least 12 IZU interventionists, must be over 18 years of age, and must be literate in Kinyarwanda.

Exclusion Criteria:

* Household exclusion criteria: Potential participants will be excluded if they do not meet the inclusion criteria above, are experiencing an active crisis (e.g., psychosis), or have severe cognitive impairments which preclude their ability to speak to the research questions/assessments under scrutiny.
* Government Official exclusion criteria: Government officials will be excluded from participation in the PLAY Collaborative if they are not located at the Cell, Sector or District level and if they are unable to meet the demands of participation in the PLAY Collaborative.
* IZU interventionist exclusion criteria: IZUs will be excluded from participation if they do not meet the inclusion criteria above and if they are unable to meet the demands of delivering the Sugira Muryango program.
* Cell Level IZU Mentor exclusion criteria: Cell Level IZU Coordinators will be excluded if they do not meet the inclusion criteria above or are unable to meet the demands of supporting the delivery of the Sugira Muryango program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1810 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Risk of Harm cases time to resolution | Through study completion, an average of 4 months
  Risk of harm cases' (violence, mental health) time to resolution in days.
Intervention Quality of Delivery | Through study completion, an average of 4 months
  Quality of delivery consists of fidelity, the ability to adhere intervention's planned activities, processes, and design, and competence, core interpersonal and professional skills relevant to mental health and psychosocial services interventions (i.e., empathy, active listening, rapport building). Fidelity is captured by intervention, session-specific items mapping planned activities and processes. Competence is capture by items mapping a set of cross-cutting interventionist skills that should be used or deployed during intervention delivery. Items are scored on a scale from 0 to 4. Scales scores are transformed and reported as percentages, with higher percentages representing higher fidelity and competence.
IZU - interventionist self-efficacy (Adapted Provider Self-efficacy scale) | Through study completion, an average of 4 months
  The Adapted Provider Self-efficacy scale measures providers' belief in ability to successfully perform specific tasks, make decisions, and deliver care. It captures confidence in the providers' skills, knowledge, and ability to manage clinical/intervention-related and interpersonal challenges effectively. Range 0-5, with higher values indicating higher self-efficacy.
John Hopkins' Dissemination and Implementation Battery (D&I) | Post-intervention, on average 4 months from baseline assessment.
  This measure is administered to interventionists, households, and organizations. It assess key implementation science domains related to buy-in, acceptability, feasibility, and appropriateness. Items are scored on a 4-point Likert scale (0-3) with higher scores indicating higher buy-in, acceptability, feasibility, etc.
The Implementation Leadership Scale (ILS) | Baseline (Pre-intervention), 4-months (Post Intervention)
  This assessment assesses a key implementation science construct regarding leadership across 4 domains (proactive leadership, knowledgeable leadership, supportive leadership, perseverant leadership). The ILS includes 12-items scored on a 5-point Likert scale (0-4) with higher scores indicating stronger leadership.
Program Sustainability Assessment Tool (PSAT) | Baseline (Pre-intervention), 4-months (Post Intervention)
  This assessment is administered to providers and organizations. It assesses sustainability of the Sugira Muryango intervention across 8 domains (environment, funding stability, partnerships, organizational capacity, program evaluation, program adaption, communication, strategic planning). The PSAT includes 40 items that are scored on a 7-point Likert scale (1-7) with higher scores indicating higher capacity for program sustainability.
Implementation Network Metrics and Characteristics | Baseline (Pre-intervention), 4-months (Post Intervention)
  Data from supervisors, IZUs, and sector-level officials will be collected using an open-ended, name-generator relational network survey. Key outcomes and metrics include network-level (size, density, reciprocity, centralization, core-periphery indices) and actor-level measures (degree, closeness, and betweenness centrality). Implementation networks graphical representations will also be compared.
Rwanda Demographic Health Survey- Intimate Partner Violence | Baseline (Pre-intervention), 4-months (Post Intervention)
  Indicators from the Rwanda DHS cover topics related to perpetration and victimization of violence between intimate partners.
Quality of Life (EQ-5D-3L) | Baseline (Pre-intervention), 4-months (Post Intervention)
  The EQ-5D-3L is a standardized, self-reported questionnaire used to measure health-related quality of life/ The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

SECONDARY OUTCOMES:
Hopkin's Symptom Checklist (HSCL) | Baseline (Pre-intervention), 4-months (Post Intervention)
  Assesses caregiver mental health including two subscales related to anxiety and depression. The HSCL includes 25 items scored on a 4-point Likert scale (1-4) scores can range from 1 to 100 with higher scores indicating poorer mental health. .
Difficulties in Emotion Regulation (DERS) | Baseline (Pre-intervention), 4-months (Post Intervention)
  Assesses caregiver emotion regulation. The full DERS scale includes 36 items which are scored on a 5-point Likert scale (1-5). Higher scores indicate greater difficulties in emotion regulation with a minimum score of 36 and maximum score of 180.
Trauma History and Post-Traumatic Stress Disorder (UCLA PTSD) | Baseline (Pre-intervention), 4-months (Post Intervention)
  Is an evidence-based tool for assessing trauma exposure and symptoms of post-traumatic stress disorder. it includes separate modules for evaluating Trauma Exposure (nature and number of potentially traumatic events experienced or witnessed) and PTSD Symptoms (symptom inventory aligned with the diagnostic criteria for PTSD as defined in the DSM. The index is structured to assess key symptom clusters, such as re-experiencing, avoidance, negative alterations in cognition and mood, and hyperarousal. Scoring helps clinicians determine symptom severity and meet diagnostic criteria for PTSD.
UNICEF MICS: Child Discipline Module | Baseline (Pre-intervention), 4-months (Post Intervention)
  A key component of the Multiple Indicator Cluster Surveys (MICS), designed by UNICEF to collect internationally comparable data on child well-being. This module captures caregivers' disciplinary practices used with children aged 1-17 years, providing insights into the prevalence of both positive and negative disciplinary methods. Assesses caregiver's disciplinary practices in three domains: Non-violent discipline, Psychological Aggression, and Physical Punishment.
Gender Equitable Men (GEM) scale | Baseline (Pre-intervention), 4-months (Post Intervention)
  Self-reported instrument that captures attitudes toward gender norms in intimate relationships or differing social expectations for men and women through two subscales: equitable and inequitable norms. The topics are on daily tasks and chores, relationships, health, and domestic violence. Scores range from 1-5 with higher scores representing higher gender equitable attitudes.
WHO infant and young child feeding practices | Baseline (Pre-intervention), 4-months (Post Intervention)
  Designed to gather information on breastfeeding and complementary feeding practices for children under the age of 2 years. This module aligns with guidelines established by the World Health Organization (WHO) to monitor child nutrition and inform programs aimed at improving feeding practices and reducing malnutrition among infants and young children. It assesses children's nutritional intake by parent-reported dietary intake reflecting the number of food groups (out of 7) the child consumed in the past 24 hours.
Observation of Caregiver-Child Interaction (OCCI) | Baseline (Pre-intervention), 4-months (Post Intervention)
  A structured observational measure designed to assess the quality of interactions between mothers (or primary caregivers) and young children (6 months - 3 years) in a natural or semi-structured setting. This tool is primarily used in research and intervention programs to examine parenting practices, early child stimulation, and responsive caregiving.
UNICEF MICS Family Care Indicators (FCI) | Baseline (Pre-intervention), 4-months (Post Intervention)
  A set of measures included in the Multiple Indicator Cluster Surveys (MICS) to assess the extent to which children are receiving adequate care, stimulation, and support for their cognitive, emotional, and social development during early childhood. The early stimulation questions are caregivers' self-reported and captures engagement in stimulating activities (e.g., reading books, playing, counting, etc.) with the child during the prior three days.

OTHER OUTCOMES:
WASH Indicators - Rwanda Demographic and Health Survey (DHS) | Baseline (Pre-intervention), 4-months (Post Intervention)
  The WASH Indicators in the Rwanda Demographic and Health Survey (DHS) refer to a set of measures designed to evaluate access to and the quality of Water, Sanitation, and Hygiene (WASH) services in households.
Ages and Stages Questionnaire-3 (ASQ-3) | Baseline (Pre-intervention), 4-months (Post Intervention)
  The ASQ uses a series of parent-completed range age-specific questionnaires designed to screen for developmental delay of children in the areas of gross motor skills, fine motor skills, communication, and problem solving. The ASQ-3 is scored using standard guidelines for standardization resulting in binary outcome variables for each domain indicating whether or not the child showed "developmental delay" vs. "no developmental delay.
Preschool Self-Regulation Assessment (PSRA) | Baseline (Pre-intervention), 4-months (Post Intervention)
  The Preschool Self-Regulation Assessment (PSRA) is a standardized tool designed to measure self-regulation skills in preschool-aged children. It is particularly used in early childhood research to assess children's emotional, attentional, and behavioral regulation abilities in structured settings. Scores range from 0 to 3, with higher scores representing higher self-regulation.
Home Observation for Measurement of the Environment (HOME) Inventory | Baseline (Pre-intervention), 4-months (Post Intervention)
  The HOME is a 43-item survey to assess psychosocial stimulation in the households and includes items on responsive caregiving, language stimulation, personal-social development, stimulation materials in the house, among others. The HOME combines observation of parenting behaviors and household conditions with caregiver report. Items are summed to derive a total score with a minimum score of 0 and a maximum score of 43. Higher home scores indicate higher levels of psychosocial stimulation in the households.
Infant Behavior Questionnaire / Early Childhood Behavior Questionnaire | Baseline (Pre-intervention), 4-months (Post Intervention)
  Caregiver report of child's temperament, on three main domains:
  (1) Surgency/Extraversion (e.g., Vocal Reactivity, High Intensity Pleasure, Smiling and Laughter, Activity Level, and Perceptual Sensitivity); (2) Negative Affectivity (Sadness, Distress to Limitations, Fear, and Falling Reactivity/Rate of Recovery from Distress) and 3) Orienting/Regulation (Low Intensity Pleasure, Cuddliness, Duration of Orienting, and Soothability).
DHS/Promundo "Father Engagement & Financial Decision-Making" survey | Baseline (Pre-intervention), 4-months (Post Intervention)
  Caregiver self-report of financial decision making and father engagement in child caretaking activities

CONTACTS AND LOCATIONS:
Overall Officials: Theresa S Betancourt, MA, Sc.D., Principal Investigator — Boston College Research Program on Children and Adversity
Locations (1):
- FXB-Rwanda / 2XHQ+F2G Umerenge wa Runda, Runda, Rwanda, Kigali, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: Yes
The study will share de-identified datasets, ensuring that all direct identifiers (DIs) are masked to protect participant confidentiality. These datasets will include relevant demographic information and outcome measures collected as part of the study. To facilitate ease of use and understanding, comprehensive codebooks and data dictionaries will also be made available, providing clear documentation of variables, coding schemes, and data definitions.
Supporting Information: Study Protocol, SAP
Time Frame: NIMH timelines and submissions schedules will be followed to share the necessary information with potential users.
Access Criteria: Study data and other relevant information will be made publicly available through the NIH National Data Archive system

REFERENCES:
- [Background] Public-Private Infrastructure Advisory Facility. Rwanda: Optimization of the KTRN national fiber backbone and 4G network. Published online April 1, 2019
- [Background] Desmond C, Watt KG, Jensen SKG, Simmons E, Murray SM, Farrar J, Placencio-Castro M, Sezibera V, Rawlings LB, Wilson B, Betancourt TS. Measuring the cost-effectiveness of a home-visiting intervention to promote early child development among rural families linked to the Rwandan social protection system. PLOS Glob Public Health. 2023 Oct 24;3(10):e0002473. doi: 10.1371/journal.pgph.0002473. eCollection 2023. PMID 37874790
- [Background] Moullin JC, Dickson KS, Stadnick NA, Rabin B, Aarons GA. Systematic review of the Exploration, Preparation, Implementation, Sustainment (EPIS) framework. Implement Sci. 2019 Jan 5;14(1):1. doi: 10.1186/s13012-018-0842-6. PMID 30611302
- [Background] Betancourt TS, Jensen SKG, Barnhart DA, Brennan RT, Murray SM, Yousafzai AK, Farrar J, Godfroid K, Bazubagira SM, Rawlings LB, Wilson B, Sezibera V, Kamurase A. Promoting parent-child relationships and preventing violence via home-visiting: a pre-post cluster randomised trial among Rwandan families linked to social protection programmes. BMC Public Health. 2020 May 6;20(1):621. doi: 10.1186/s12889-020-08693-7. PMID 32375840
- [Background] Aarons GA, Fettes DL, Hurlburt MS, Palinkas LA, Gunderson L, Willging CE, Chaffin MJ. Collaboration, negotiation, and coalescence for interagency-collaborative teams to scale-up evidence-based practice. J Clin Child Adolesc Psychol. 2014;43(6):915-28. doi: 10.1080/15374416.2013.876642. Epub 2014 Mar 10. PMID 24611580
- [Background] Aarons GA, Hurlburt M, Horwitz SM. Advancing a conceptual model of evidence-based practice implementation in public service sectors. Adm Policy Ment Health. 2011 Jan;38(1):4-23. doi: 10.1007/s10488-010-0327-7. PMID 21197565
- [Background] Jensen SK, Placencio-Castro M, Murray SM, Brennan RT, Goshev S, Farrar J, Yousafzai A, Rawlings LB, Wilson B, Habyarimana E, Sezibera V, Betancourt TS. Effect of a home-visiting parenting program to promote early childhood development and prevent violence: a cluster-randomized trial in Rwanda. BMJ Glob Health. 2021 Jan;6(1):e003508. doi: 10.1136/bmjgh-2020-003508. PMID 33514591
- [Background] Betancourt TS, Thomson D, VanderWeele TJ. War-Related Traumas and Mental Health Across Generations. JAMA Psychiatry. 2018 Jan 1;75(1):5-6. doi: 10.1001/jamapsychiatry.2017.3530. No abstract available. PMID 29188290
- [Background] Jensen SKG, Sezibera V, Murray SM, Brennan RT, Betancourt TS. Intergenerational impacts of trauma and hardship through parenting. J Child Psychol Psychiatry. 2021 Aug;62(8):989-999. doi: 10.1111/jcpp.13359. Epub 2020 Dec 7. PMID 33284991
- [Background] Betancourt TS, Williams TP, Kellner SE, Gebre-Medhin J, Hann K, Kayiteshonga Y. Interrelatedness of child health, protection and well-being: an application of the SAFE model in Rwanda. Soc Sci Med. 2012 May;74(10):1504-11. doi: 10.1016/j.socscimed.2012.01.030. Epub 2012 Mar 9. PMID 22459187
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052